CLINICAL TRIAL: NCT05688878
Title: Patient Experiences With Threshold Electrical Stimulation İn Stroke: A Qualitative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qualitative study about TES
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: stroke; electric stimulation; qualitative research; sensory thresholds
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: An exploratory-descriptive qualitative study will be conducted . This study will be conducted with 10 stroke patients receiving threshold electrical stimulation therapy. Threshold electrical stimulation will be applied for 4 weeks, 3 days a week, for one hour. At the end of the 4th week, semi-structured focus group interviews will be held with the patients. . In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Compared to taking notes by hand; It will be preferable to record the conversation with a voice recorder because it has advantages such as recording all the interviews and allowing the interviewer to focus on the interview. Thematic analysis method will be used in the evaluation of the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): An exploratory-descriptive qualitative study will be conducted . This study will be conducted with 10 stroke patients receiving threshold electrical stimulation therapy. Threshold electrical stimulation will be applied for 4 weeks, 3 days a week, for one hour. At the end of the 4th week, semi-structured focus group interviews will be held with the patients. . In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Compared to taking notes by hand; It will be preferable to record the conversation with a voice recorder because it has advantages such as recording all the interviews and allowing the interviewer to focus on the interview. Thematic analysis method will be used in the evaluation of the data.
  Interventions: Device: Threshold electrical stimulation

INTERVENTIONS:
Device: Threshold electrical stimulation — Threshold stimulation (EDS) is based on low-intensity (<100 Hz) and long-duration current and is applied with superficial electrodes. Threshold stimulation provides a natural proprioception by depolarizing the sensory and motor nerves without causing any muscle contraction.This treatment will be applied for 4 weeks, 3 days a week, for 1 hour.

SUMMARY:
The aim of this study is to determine patient opinions and experiences about threshold electrical stimulation treatment applied to stroke patients.

DETAILED DESCRIPTION:
An exploratory-descriptive qualitative study will be conducted . This study will be conducted with 10 stroke patients receiving threshold electrical stimulation therapy. Threshold electrical stimulation will be applied for 4 weeks, 3 days a week, for one hour. At the end of the 4th week, semi-structured focus group interviews will be held with the patients. . In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Compared to taking notes by hand; It will be preferable to record the conversation with a voice recorder because it has advantages such as recording all the interviews and allowing the interviewer to focus on the interview. Thematic analysis method will be used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 80 years,
* Individuals without communication problems,
* Individuals who have been diagnosed with stroke

Exclusion Criteria:

* Uncontrollable arrhythmia and/or hypertension
* Presence of advanced sensory deficit
* Visual and hearing problems
* Not having sufficient communication skills (Mini Mental Test score below 24 points)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Semi-structured focus group interviews about patients' Perception of threshold electrical stimulation | Change from baseline Patients' Perception of Threshold electrical stimulation at week 4
  At the end of the 4th week, semi-structured focus group interviews will be held with the patients. . In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Thematic analysis method will be used in the evaluation of the data

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided